CLINICAL TRIAL: NCT02648152
Title: Multicenter Clinical Observation Using the Cementless Version of the POLARSTEM
Brief Title: POLARSTEM Cementless Hip Stem
Acronym: POLARSTEM
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D10070-1
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2021-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Total Hip Arthroplasty — Total Hip Arthroplasty using Cementless version of the POLARSTEM

SUMMARY:
Multicenter observational study to validate that the POLARSTEM™ is a state-of-the-art implant in terms of radiographic, clinical performance and long-term survivorship.

DETAILED DESCRIPTION:
The goal of this multicenter clinical observation is to validate short-, mid-, and long-term outcome (efficacy and safety) of the POLARSTEM™.

Efficacy evaluations:

* Evaluation of function, range of motion (ROM) and pain as assessed by Harris Hip Score, Hip disability and osteoarthritis outcome score (HOOS) [7, 8], an extension of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
* Radiographic changes as defined by radiolucent lines, osteolysis, hypo- and hypertrophy, implant loosening or migration

Safety evaluations:

* Intra- and perioperative device-related adverse events (AE) and complications up to discharge
* Postoperative AE up to 10 years

ELIGIBILITY:
Inclusion Criteria:

* Patient has no general medical contraindication to surgery
* Informed consent to participate in the MCO signed by the patient
* Routine radiographic assessment is possible
* Patient is likely to comply with study follow-up requirements
* Primary total hip replacement (THR) to the affected side, unilateral or bilateral

Exclusion Criteria:

* Previously failed endoprosthesis and /or THR components in relevant hip
* History of infection in the affected joint; systemic infections
* Grossly insufficient femoral or acetabular bone stock in the involved hip
* Charcot joint disease or other severe neurosensory deficit
* Severe spinal disorders
* Age of patient at date of surgery > 75 years
* High comorbidity
* Cemented acetabular cup

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this multicenter clinical observation will have at least one of the indications listed below and meet all of the inclusion criteria. Patients meeting any of the exclusion criteria are not eligible for this study.
  Indications
  * Primary or secondary coxarthrosis
  * Rheumatoid arthritis
  * Developmental dysplasia of the hip (Crowe type I and II)
  * Fracture or avascular necrosis of the femoral head
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Turgay Efe, Dr.med., Principal Investigator — Philipps University Marburg
Locations (3):
- Germany (2):
  - St. Elisabeth Hospital, Orthopedics and Rheumatology, Bochum
  - University Marburg, Orthopedics and Rheumatology, Marburg
- Kantonsspital Aarau, Orthopedics, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cypres A, Fiquet A, Girardin P, Fitch D, Bauchu P, Bonnard O, Noyer D, Roy C. Long-term outcomes of a dual-mobility cup and cementless triple-taper femoral stem combination in total hip replacement: a multicenter retrospective analysis. J Orthop Surg Res. 2019 Nov 21;14(1):376. doi: 10.1186/s13018-019-1436-y. PMID 31752951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at three centers in two countries in Europe (2 in Germany and 1 in Switzerland)
Units Other Than Participants: hips
Period: Overall Study
Arm/Group | Total Hip Arthroplasty
Started | 218; 225 hips
Completed | 94; 96 hips (Site: Chefarzt Orthopädische Klinik stopped participation in the study prior to study completion at the 10 year follow-up point. The decision was made by the site due to the institution reducing staff.)
Not Completed | 124; 129 hips

BASELINE CHARACTERISTICS:
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.70 (7.70)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <= 60 years | 62
  Age Group: > 60 years | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.30 (4.72)

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate: Overall Survivorship of POLARSTEM
Description: Overall survivorship of the Cementless Version of the POLARSTEM pre-operatively, 3 months, 12 months, 12 months, 36 months, 60 months, and 120 months by Kaplan-Meier estimate with overall hip survivorship defined as the time between date of treatment and date of revision for any reason.
Time Frame: Pre-operatively, 3 months, 12 months, 36 months, 60 months, and 120 months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Number (95% Confidence Interval); unit: percentage of hips
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
percentage of hips
  Pre-operatively | 100 — Lower and Upper 95% Confidence Interval limit not estimable for baseline (pre-operative) time point.
  3 Months: number analyzed (Participants) | 217
  3 Months: number analyzed (hips) | 224
  3 Months | 99.6 [96.9 to 99.9]
  12 Months: number analyzed (Participants) | 215
  12 Months: number analyzed (hips) | 222
  12 Months | 99.1 [96.5 to 99.8]
  36 Months: number analyzed (Participants) | 212
  36 Months: number analyzed (hips) | 219
  36 Months | 98.7 [95.9 to 99.6]
  60 Months: number analyzed (Participants) | 170
  60 Months: number analyzed (hips) | 174
  60 Months | 98.7 [95.9 to 99.6]
  120 Months: number analyzed (Participants) | 132
  120 Months: number analyzed (hips) | 133
  120 Months | 98.7 [95.9 to 99.6]

2. Secondary Outcome: Harris Hip Score (HHS)
Description: The HHS measured function, range of motion (ROM), and pain sub-scores that are combined to indicate total dysfunction on a numerical scale from 0 to 100, with a higher score indicating less dysfunction (i.e., a better outcome). Reported scores for the HHS utilized the following grading:
  * <70 = poor
  * 70 to 80 = fair
  * 80 to 90 = good
  * 90 to 100 = excellent
Time Frame: Pre-operative, 3 Months, 12 Months, 36 Months, 60 Months, 120 months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
score on a scale
  Pre-operative | 48.60 (11.55)
  3 Months: number analyzed (Participants) | 207
  3 Months: number analyzed (hips) | 214
  3 Months | 83.10 (13.24)
  12 Months: number analyzed (Participants) | 210
  12 Months: number analyzed (hips) | 217
  12 Months | 89.20 (12.71)
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 191
  36 Months | 89.10 (13.06)
  60 Months: number analyzed (Participants) | 161
  60 Months: number analyzed (hips) | 166
  60 Months | 88.00 (15.24)
  120 Months: number analyzed (Participants) | 62
  120 Months: number analyzed (hips) | 63
  120 Months | 85.30 (14.92)

3. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): Pain Subscale
Description: WOMAC Pain subscale is a subset of the Hip Disability and Osteoarthritis Outcome Score (HOOS) with a range of 0 to 20. Higher WOMAC scores indicate worse pain (i.e., worse outcome) and lower scores indicate less pain (i.e., a better outcome).
Time Frame: Pre-operative, 3 Months, 12 Months, 36 Months, 60 Months, 120 Months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
score on a scale
  Pre-operative | 11.5 (3.08)
  3 Months: number analyzed (Participants) | 208
  3 Months: number analyzed (hips) | 215
  3 Months | 1.9 (2.46)
  12 Months: number analyzed (Participants) | 210
  12 Months: number analyzed (hips) | 217
  12 Months | 1.5 (2.21)
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 191
  36 Months | 1.7 (2.64)
  60 Months: number analyzed (Participants) | 175
  60 Months: number analyzed (hips) | 180
  60 Months | 1.5 (2.75)
  120 Months: number analyzed (Participants) | 94
  120 Months: number analyzed (hips) | 96
  120 Months | 1.0 (2.46)

4. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): Stiffness Subscale
Description: WOMAC Stiffness subscale is a subset of the Hip Disability and Osteoarthritis Outcome Score (HOOS) with a range from 0 to 8 with a higher score indicating a worse outcome and a low score indicating a better outcome.
Time Frame: Pre-operative, 3 Months, 12 Months, 36 Months, 60 Months, 120 Months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
score on a scale
  Pre-operative | 5.0 (1.46)
  3 Months: number analyzed (Participants) | 208
  3 Months: number analyzed (hips) | 215
  3 Months | 1.6 (1.50)
  12 Months: number analyzed (Participants) | 210
  12 Months: number analyzed (hips) | 217
  12 Months | 1.1 (1.24)
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 191
  36 Months | 1.0 (1.51)
  60 Months: number analyzed (Participants) | 175
  60 Months: number analyzed (hips) | 180
  60 Months | 0.7 (1.24)
  120 Months: number analyzed (Participants) | 94
  120 Months: number analyzed (hips) | 96
  120 Months | 0.6 (1.22)

5. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): Physical Function Subscale
Description: WOMAC Physical Function subscale is a subset of the Hip Disability and Osteoarthritis Outcome Score (HOOS) with a range from 0 to 68 with a higher score indicating a worse outcome and a low score indicating a better outcome.
Time Frame: Pre-operative, 3 Months, 12 Months, 36 Months, 60 Months, 120 Months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
score on a scale
  Pre-operative | 42.1 (10.53)
  3 Months: number analyzed (Participants) | 208
  3 Months: number analyzed (hips) | 215
  3 Months | 10.8 (11.21)
  12 Months: number analyzed (Participants) | 210
  12 Months: number analyzed (hips) | 217
  12 Months | 8.0 (9.42)
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 191
  36 Months | 8.0 (11.23)
  60 Months: number analyzed (Participants) | 175
  60 Months: number analyzed (hips) | 180
  60 Months | 9.3 (11.35)
  120 Months: number analyzed (Participants) | 94
  120 Months: number analyzed (hips) | 96
  120 Months | 5.9 (10.10)

6. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): Total Score
Description: WOMAC total score combines Stiffness, Pain, and Physical Function subscales of the Hip Disability and Osteoarthritis Outcome Score (HOOS) into a range from 0 to 96 with a higher score indicating a worse outcome and a lower score indicating a better outcome.
Time Frame: Pre-operative, 3 Months, 12 Months, 36 Months, 60 Months, 120 Months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 218
Number analyzed (hips) | 225
score on a scale
  Pre-operative | 58.6 (13.94)
  3 Months: number analyzed (Participants) | 208
  3 Months: number analyzed (hips) | 215
  3 Months | 14.2 (14.39)
  12 Months: number analyzed (Participants) | 210
  12 Months: number analyzed (hips) | 217
  12 Months | 10.5 (12.11)
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 191
  36 Months | 10.7 (14.53)
  60 Months: number analyzed (Participants) | 175
  60 Months: number analyzed (hips) | 180
  60 Months | 11.6 (14.38)
  120 Months: number analyzed (Participants) | 94
  120 Months: number analyzed (hips) | 96
  120 Months | 7.4 (12.91)

7. Secondary Outcome: Radiological: Radiolucent Lines
Description: Number of hips identified with radiographic findings of radiolucent lines present (Yes/No) in femoral zones 1 to 14. Radiolucent lines indicated seams of 0 millimeters to 2 millimeters or greater.
Time Frame: 3 months, 12 months, 36 months, 60 months, 120 months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 212
Number analyzed (hips) | 219
hips
  3 Months: Yes | 2
  3 Months: No | 217
  12 Months: number analyzed (Participants) | 208
  12 Months: number analyzed (hips) | 215
  12 Months: Yes | 0
  12 Months: No | 215
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 190
  36 Months: Yes | 7
  36 Months: No | 183
  60 Months: number analyzed (Participants) | 161
  60 Months: number analyzed (hips) | 166
  60 Months: Yes | 1
  60 Months: No | 165
  120 Months: number analyzed (Participants) | 63
  120 Months: number analyzed (hips) | 64
  120 Months: Yes | 2
  120 Months: No | 62

8. Secondary Outcome: Radiological: Osteolysis
Description: Number of hips identified with radiographic findings of osteolysis present (Yes/No) in femoral zones 1 to 14.
Time Frame: 3 months, 12 months, 36 months, 60 months, 120 months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 212
Number analyzed (hips) | 219
hips
  3 Months: Yes | 0
  3 Months: No | 219
  12 Months: number analyzed (Participants) | 208
  12 Months: number analyzed (hips) | 215
  12 Months: Yes | 1
  12 Months: No | 214
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 190
  36 Months: Yes | 1
  36 Months: No | 189
  60 Months: number analyzed (Participants) | 161
  60 Months: number analyzed (hips) | 166
  60 Months: Yes | 0
  60 Months: No | 166
  120 Months: number analyzed (Participants) | 63
  120 Months: number analyzed (hips) | 64
  120 Months: Yes | 3
  120 Months: No | 61

9. Secondary Outcome: Radiological: Atrophy
Description: Number of hips identified with radiographic findings for atrophy in femoral zones 1 to 14 indicated as:
  * None
  * Mild
  * Moderate
  * Severe
  * Missing
Time Frame: 3 months, 12 months, 36 months, 60 months, 120 months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 212
Number analyzed (hips) | 219
hips
  3 Months: None | 1
  3 Months: Mild | 0
  3 Months: Moderate | 0
  3 Months: Severe | 0
  3 Months: Missing | 218
  12 Months: number analyzed (Participants) | 208
  12 Months: number analyzed (hips) | 215
  12 Months: None | 0
  12 Months: Mild | 0
  12 Months: Moderate | 0
  12 Months: Severe | 0
  12 Months: Missing | 215
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 190
  36 Months: None | 1
  36 Months: Mild | 0
  36 Months: Moderate | 0
  36 Months: Severe | 0
  36 Months: Missing | 189
  60 Months: number analyzed (Participants) | 161
  60 Months: number analyzed (hips) | 166
  60 Months: None | 0
  60 Months: Mild | 1
  60 Months: Moderate | 0
  60 Months: Severe | 0
  60 Months: Missing | 165
  120 Months: number analyzed (Participants) | 63
  120 Months: number analyzed (hips) | 64
  120 Months: None | 0
  120 Months: Mild | 0
  120 Months: Moderate | 0
  120 Months: Severe | 1
  120 Months: Missing | 63

10. Secondary Outcome: Radiological: Hypertrophy
Description: Number of hips identified with radiographic findings for hypertrophy in femoral zones 1 to 14 indicated as:
  * None
  * Mild
  * Moderate
  * Severe
  * Missing
Time Frame: 3 months, 12 months, 36 months, 60 months, 120 months
Population: All participants who received study treatment with data collected for the given outcome at the time point specified.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 212
Number analyzed (hips) | 219
hips
  3 Months: None | 0
  3 Months: Mild | 0
  3 Months: Moderate | 0
  3 Months: Severe | 0
  3 Months: Missing | 219
  12 Months: number analyzed (Participants) | 208
  12 Months: number analyzed (hips) | 215
  12 Months: None | 0
  12 Months: Mild | 0
  12 Months: Moderate | 0
  12 Months: Severe | 1
  12 Months: Missing | 214
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 190
  36 Months: None | 1
  36 Months: Mild | 0
  36 Months: Moderate | 0
  36 Months: Severe | 1
  36 Months: Missing | 188
  60 Months: number analyzed (Participants) | 161
  60 Months: number analyzed (hips) | 166
  60 Months: None | 0
  60 Months: Mild | 1
  60 Months: Moderate | 0
  60 Months: Severe | 2
  60 Months: Missing | 163
  120 Months: number analyzed (Participants) | 63
  120 Months: number analyzed (hips) | 64
  120 Months: None | 0
  120 Months: Mild | 1
  120 Months: Moderate | 0
  120 Months: Severe | 0
  120 Months: Missing | 63

11. Secondary Outcome: Radiological: Loosening of the Implant or Migration
Description: Number of hips identified with radiographic findings associated with loosening of the implant or migration were indicated as:
  * Integration not assessable
  * Indifferent, bone unchanged
  * Osteointegration, integration
  * Bone loss
  * Signs of loosening
  * Revision indicated
Time Frame: 3 months, 12 months, 36 months, 60 months, 120 months
Population: All participants who received study treatment with data available for the given outcome at the time point specified.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Total Hip Arthroplasty
Number analyzed (Participants) | 212
Number analyzed (hips) | 219
hips
  3 Months: Integration not assessable | 4
  3 Months: Indifferent, bone unchanged | 138
  3 Months: Osteointegration, integration | 77
  3 Months: Bone loss | 0
  3 Months: Signs of loosening | 0
  3 Months: Revision indicated | 0
  12 Months: number analyzed (Participants) | 208
  12 Months: number analyzed (hips) | 215
  12 Months: Integration not assessable | 0
  12 Months: Indifferent, bone unchanged | 81
  12 Months: Osteointegration, integration | 134
  12 Months: Bone loss | 0
  12 Months: Signs of loosening | 0
  12 Months: Revision indicated | 0
  36 Months: number analyzed (Participants) | 184
  36 Months: number analyzed (hips) | 190
  36 Months: Integration not assessable | 0
  36 Months: Indifferent, bone unchanged | 67
  36 Months: Osteointegration, integration | 123
  36 Months: Bone loss | 0
  36 Months: Signs of loosening | 0
  36 Months: Revision indicated | 0
  60 Months: number analyzed (Participants) | 161
  60 Months: number analyzed (hips) | 166
  60 Months: Integration not assessable | 0
  60 Months: Indifferent, bone unchanged | 104
  60 Months: Osteointegration, integration | 62
  60 Months: Bone loss | 0
  60 Months: Signs of loosening | 0
  60 Months: Revision indicated | 0
  120 Months: number analyzed (Participants) | 63
  120 Months: number analyzed (hips) | 64
  120 Months: Integration not assessable | 0
  120 Months: Indifferent, bone unchanged | 22
  120 Months: Osteointegration, integration | 40
  120 Months: Bone loss | 2
  120 Months: Signs of loosening | 0
  120 Months: Revision indicated | 0

ADVERSE EVENTS:
Time Frame: Surgery to End of Study visit, approximately 120 months
Arm/Group | Total Hip Arthroplasty
All-Cause Mortality (participants affected / at risk) | 29/218
Serious Adverse Events (participants affected / at risk) | 114/218
Other Adverse Events (participants affected / at risk) | 115/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Hip Arthroplasty (N=218)
Quadruple Heart bypass (Cardiac disorders) | 1 (1)
Abdominal Surgery due to Bridenileus - no relationship to study device (Gastrointestinal disorders) | 1 (1)
Poor general condition (General disorders) | 1 (1) — Poor general condition, especially due to COPD. Pain in the hip, which decreased after weight loss of 35kg.
ACI stenosis on both sides (Cardiac disorders) | 1 (1)
Additional abdominal surgery due to adhesions (Gastrointestinal disorders) | 1 (2)
Amputation of the small toe on the right due to melanoma (Skin and subcutaneous tissue disorders) | 1 (1)
Ankle arthrodesis on the right (Musculoskeletal and connective tissue disorders) | 1 (1)
Apoplexy (Nervous system disorders) | 1 (1)
Articulated flat splayfoot on the left, insoles adapted (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
AV fistula after cardiac catheter right groin (Cardiac disorders) | 1 (1)
Bladder cancer (Renal and urinary disorders) | 1 (1)
Breakage of inlay due to recurrent falls due to M. Parkinson (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cage-implantation L3/L4 (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract surgery on both sides (Eye disorders) | 1 (1)
Cervical spine surgery 2017 (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholecystectomy (Gastrointestinal disorders) | 2 (2)
Chronic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic kidney insufficiency (Renal and urinary disorders) | 1 (1)
Chronic renal failure (Renal and urinary disorders) | 1 (1)
Colon tumour (Gastrointestinal disorders) | 1 (1)
Condition after herniated cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Condition after herniated disc LWK1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Condition after knee TEP on the left (no complaints currently) (Musculoskeletal and connective tissue disorders) | 1 (1)
Contralateral hip TEP (Musculoskeletal and connective tissue disorders) | 1 (1)
Contralateral Hip treated with TEP to explain LLD 8mm (Musculoskeletal and connective tissue disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Coronary 2-vessel disease PAVK II bilateral (Cardiac disorders) | 1 (1)
Coronary Heart Disease (Cardiac disorders) | 2 (2)
Coronary stent (Cardiac disorders) | 2 (2)
Cup fixation (Musculoskeletal and connective tissue disorders) | 1 (1)
Cup revision after dislocation (Musculoskeletal and connective tissue disorders) | 1 (1)
Death (General disorders) | 3 (3)
Death - Death not caused or contributed to misuse of the study device (General disorders) | 1 (1)
Death due to abdominal surgery (Gastrointestinal disorders) | 1 (1)
Death due to cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death due to cardiac failure (Cardiac disorders) | 1 (1)
Death due to cervic carcinoma (Reproductive system and breast disorders) | 1 (1)
Death due to multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death due to old age - no relationship to study device (General disorders) | 1 (1)
Death due to pancreatic cancer (Hepatobiliary disorders) | 1 (1)
Death due to suicide (Psychiatric disorders) | 1 (1)
Death due to traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Death -Exitus letalis for pulmonary bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death, cause not related to hip surgery (General disorders) | 1 (1)
Death. Cause of death and information about prosthesis are not available (General disorders) | 1 (1)
Death. Cause of death is unknown (General disorders) | 1 (1)
Death. Cause of death unknown. Polarstem in situ. (General disorders) | 1 (1)
Death. Not related to hip surgery (General disorders) | 2 (2)
Death. Not related to the study procedure. The cause of death is unknown (General disorders) | 1 (1)
Death. Polarstem in situ. Cause of death unknown (General disorders) | 1 (1)
Death. Reason unknown (General disorders) | 1 (1)
Death. Reason unknown. Prosthesis in situ. (General disorders) | 1 (1)
Death: ARDS, no relation to study process visible (Respiratory, thoracic and mediastinal disorders) | 1 (1) — exitus letalis: Acute Respiratory Distress Syndrome (ARDS) after bilateral pneumonia. No relation to study process visible
Death: Hip in situ. Cause of death is unknown (General disorders) | 1 (1)
Death: Hip in situ. No further information available on the cause of death (General disorders) | 1 (1)
Death: stroke (Nervous system disorders) | 1 (1)
Deep vein thrombosis and subarachnoid haemorrhagic bleeding (Blood and lymphatic system disorders) | 1 (1)
Degenerative thoracic spine syndrome (secondary diagnosis documented) (Musculoskeletal and connective tissue disorders) | 1 (1)
Diabetes (Endocrine disorders) | 1 (1)
Diabetes (secondary diagnosis documented) (Endocrine disorders) | 1 (1)
Diabetes II (Endocrine disorders) | 2 (2)
Diabetes mellitus (Endocrine disorders) | 1 (1)
Diabetic mellitus with polyneuropathy (Endocrine disorders) | 1 (1)
Disclocation closed reposition (Musculoskeletal and connective tissue disorders) | 1 (1)
Dislocation (Luxation) (Musculoskeletal and connective tissue disorders) | 1 (1) — Dislocation of study hip connected to everyday movements. No revision or surgery due to astric ED adenocarcinoma and urgent therapy of carcinoma
Early infection (Infections and infestations) | 1 (1)
Early infection, septic revision (Musculoskeletal and connective tissue disorders) | 1 (1)
Erysipelas right lower leg (Infections and infestations) | 1 (1)
Excision of leukoplakia right soft palate (Gastrointestinal disorders) | 1 (1)
Exitus letalis: eCPR due to cardiac arrest (Cardiac disorders) | 1 (1) — Exitus letalis: eCPR due to cardiac arrest. In general no relation to study procedure. Died with hip in situ.
Foot surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot surgery hallux valgus left - no relationship to study device (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture and WK replacement C5 in 2012. Fracture C6/7 in 1997 (Musculoskeletal and connective tissue disorders) | 1 (1)
Gait disturbance most likely due to normal pressure hydrocephalus (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain, unclear aetiology left hip without organic cause (Musculoskeletal and connective tissue disorders) | 1 (1)
Heart attack (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hemiparesis right leg with force grade 4/5. (Nervous system disorders) | 1 (1)
Hip prosthesis left (Musculoskeletal and connective tissue disorders) | 5 (5)
Hip prosthesis right (opposite side) no relationship to study device (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip replacement right (Musculoskeletal and connective tissue disorders) | 6 (6)
Hip TEP (Musculoskeletal and connective tissue disorders) | 2 (2)
Hip TEP contralateral side, left, , age-related not related to study hip. (Musculoskeletal and connective tissue disorders) | 4 (4)
Hip TEP left, Implantation due to coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Normal peri and post operative progress, no relation to study process
Hip TEP. Non-study hip. Age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
HKB crack right 08'18. No association to the study procedure. (Musculoskeletal and connective tissue disorders) | 1 (1)
Hospitalisation (General disorders) | 3 (3)
Hospitalisation due to Bronchitis and Cholezystolithiasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalisation due to chronic low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hospitalisation for Artial Fibrillation (Cardiac disorders) | 1 (1)
Hospitalisation. Inpatient due to acute psychosis (Psychiatric disorders) | 1 (1)
Hospitalisation: infection after knee TP (Infections and infestations) | 1 (1)
Hospitalised for myocardial infarction (Cardiac disorders) | 1 (1)
Humerus subcapital fracture, no visible connection to study procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
Hysterectomy (Reproductive system and breast disorders) | 1 (1)
Hystorectomy. No association to the study procedure. (Reproductive system and breast disorders) | 1 (1)
Implantation of hip replacement surgery Li (Musculoskeletal and connective tissue disorders) | 1 (1)
Implantation of neurostimulator in lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Inlay loosening, malfixation during surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Inpatient conservative therapy in a hospital (General disorders) | 1 (1)
Inpatient geriatric for asthma, no relationship to study device (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inpatient geriatric for dementia, no relationship to study device (Psychiatric disorders) | 1 (1)
Intervetebral disc surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Intestinal Obstruction (Ileus) with adhesions with surgery (Gastrointestinal disorders) | 1 (1)
July 2019 facet joint surgery spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee prosthesis right (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee replacement - left (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee replacement - right (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP bilateral (date unknown), age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP both sides (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP due to progressive pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP left (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP on both sides (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP right (Musculoskeletal and connective tissue disorders) | 5 (6)
Knee TEP right date unknown, age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP right due to gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP right side (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP right side, date unknown, not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP right. Age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee total replacement left (Musculoskeletal and connective tissue disorders) | 1 (1)
Left gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip prosthesis (non-study hip) (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip TEP (non-study hip) (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip TEP, Primary coxarthroses (Musculoskeletal and connective tissue disorders) | 1 (1) — Normal peri and post operative progress. No visible relation to study procedure.
Leg length difference compensated accoridng to patient information (Musculoskeletal and connective tissue disorders) | 1 (1)
Length discrepancy corrected with shoe insole (Musculoskeletal and connective tissue disorders) | 1 (1)
Local infection (Infections and infestations) | 1 (1)
Long biceps tendon tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung embolism after study procedure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Mammary carcinoma (Reproductive system and breast disorders) | 1 (1)
Massive pain due to functional limitation of non study hip (Coxarthrose contralateral side) (Musculoskeletal and connective tissue disorders) | 1 (1)
Mental problems (Psychiatric disorders) | 1 (1)
Metastasis liver (Hepatobiliary disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Numbness since surgery in 4.and 5. toe and outer side of the left foot. (Nervous system disorders) | 1 (1)
Operation in esophagus CA (Gastrointestinal disorders) | 1 (1)
Opiate and benzodiazepine addiction (Psychiatric disorders) | 1 (1)
OSAS with CPAP (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Osteoarthritis left knee, right hip. No association with the study process visible (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain after stent surgery in the area of arteria iliaca externa (Cardiac disorders) | 1 (1)
Bronchial cancer (NSCLC) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchial cancer (NSCLC) first diagnosis 2011 with metastasis resection of parietal lobes 12/2013 and 11/2014. Parietal lobe resection surgery due to lung cancer
Perforated stomach ulcer (malign) (Gastrointestinal disorders) | 1 (1)
Peripheral artery disease bilateral with percutaneous transluminal angioplasty (PTA) left (Cardiac disorders) | 1 (1)
Periprosthetic femoral fracture left (Musculoskeletal and connective tissue disorders) | 1 (1)
Peroneus partial palsy left (Nervous system disorders) | 1 (1)
Pleural effusion Jan 2016, Pleurodesis 15.06.2016 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polineuropathy (Nervous system disorders) | 1 (1)
Possible trochanteric fracture after a fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Postoperative failure of kidney implant. High Crea 3,3mg/dl (Renal and urinary disorders) | 1 (1)
Prostate cancer (Renal and urinary disorders) | 1 (1)
Proximal high grade stenosis in tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Radial fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Removal of haematoma after falling right thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Re-operation head change and inlay change (Musculoskeletal and connective tissue disorders) | 1 (1)
Restriction due to spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Right forearm fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Right knee TEP, with complaints (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff rupture on both sides - no evidence of a connection with study procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p cataract surgery (Eye disorders) | 1 (1)
s/p detached retina with eye surgery (Eye disorders) | 1 (1)
s/p disc prolapse surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p disc prolapse surgery. No relation to study procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p fracture of the shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p hip TEP left (Musculoskeletal and connective tissue disorders) | 2 (2)
Secretion in liver (Hepatobiliary disorders) | 1 (1)
Semantic dementia first diagnosis (Psychiatric disorders) | 1 (1)
Shoulder surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder surgery, partial rotator cuff rupture right (Musculoskeletal and connective tissue disorders) | 1 (1) — Degenerative rupture of the long biceps tendon right. No relation to the study procedure visible
Shoulder TEP, left side, date unknown, not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder TEP. Not related to study procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
Shunt implantation for normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Sintering fracture of a lumbar vertebra (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal surgery after a herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Spine/inpation treatment for lumbar disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylectomy L1-S1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Steatosis hepatis (Hepatobiliary disorders) | 1 (1)
Suspected fissural tibial shaft fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
THA left (non-study hip) (Musculoskeletal and connective tissue disorders) | 1 (1)
Thoracic spine fracture (BWS-12), traumatic brain injury (Musculoskeletal and connective tissue disorders) | 1 (1) — Avulsion of the extensor digitorum in fingers, sternal fracture, rib fracture, subdural haematoma
Three-vessel disease (Cardiac disorders) | 1 (1)
Thyroid carcinoma. No association with the study process visible (Endocrine disorders) | 1 (1)
TIA left hemisphere (Nervous system disorders) | 1 (1)
TKA (Musculoskeletal and connective tissue disorders) | 1 (1)
Total hip replacement on left side (Musculoskeletal and connective tissue disorders) | 1 (1)
Type 2 diabetes mellitus (Endocrine disorders) | 1 (1)
Ulnar and radius fracture. Pre-existing condition (Musculoskeletal and connective tissue disorders) | 1 (1)
Varicosis OP. No association with the study process visible (Cardiac disorders) | 1 (1)
VHF arterial fibrillation (medication) (Cardiac disorders) | 1 (1)
Walking affected due to hip TEP on both sides (Musculoskeletal and connective tissue disorders) | 1 (1) — Hip TEP opposite side date unknown, age-related, not related to study hip
Z. n. Pancreas cancer (Hepatobiliary disorders) | 1 (1)
Z.n. acute kidney failure (Renal and urinary disorders) | 1 (1)
Z.n. bypass right leg (Cardiac disorders) | 1 (1)
Z.n. decompression lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Z.n. herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Z.n. Pneumonia bilateral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Z.n. Pulmonary embolism with thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Z.n.TBVT li (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Hip Arthroplasty (N=218)
Absolute arrhythmia atrial fibrillation (Cardiac disorders) | 1 (1)
Addiction syndrom (Psychiatric disorders) | 1 (1)
Advanced right coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aortic insufficiency (Cardiac disorders) | 1 (1)
Aortic stenosis (Cardiac disorders) | 1 (1)
Arterial hypertension (Cardiac disorders) | 8 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis in feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthrosis left knee (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthrosis left talocrural joint (OSG) no surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrosis LWK 4 & 5 (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrosis. No relation to study procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Back pain due to obesity and age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder catheter (Renal and urinary disorders) | 1 (1)
Bleeding tendency (blood loss 1.5L) (Blood and lymphatic system disorders) | 1 (1)
Bronchial asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruised ribs (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis trochanterica (Musculoskeletal and connective tissue disorders) | 1 (1)
Can walk stairs and ascents very poorly due to muscular insufficiency. Avoids standing for long time (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac insufficiency (Cardiac disorders) | 1 (1)
Cardiovascular disturbances (Cardiac disorders) | 5 (5)
Cholecystolithiasis (not related to study procedure) (Gastrointestinal disorders) | 1 (1)
Chronic gastric ulcer (Gastrointestinal disorders) | 1 (1)
Condition after bursitis of the thighs on both sides (Musculoskeletal and connective tissue disorders) | 1 (1)
COPD with continuous oxygen administration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary heart disease (Cardiac disorders) | 2 (2)
Coxarthrosis on the left, SIG arthrosis on both sides (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramp-like pain on prolonged exposure in the lateral thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Decubitus Heel (Musculoskeletal and connective tissue disorders) | 1 (1)
Demolition d. major trochanter tip in the process of being resorbed (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diabetis mellitus regulation disorder (Endocrine disorders) | 1 (1)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disc prolapse cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Disc prolapse in lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Disc prolapse in the L4/L5 area (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Early complications: pressure ulcers. 1st degree on the sacrum (Skin and subcutaneous tissue disorders) | 1 (1)
Extreme knee and back pain. Condition after a five-fold herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall on both hips ~3 months ago (Musculoskeletal and connective tissue disorders) | 1 (1) — Additionally complaints in the area of lumbar spine and in the area of the SI joint with severe pressure pain
Fall on the hip twice (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall. Stabbing groin pain since then (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastritis (not related to study procedure) (Gastrointestinal disorders) | 1 (1)
GIST des sigmas with sigma resection (Gastrointestinal disorders) | 1 (1)
Gluteal muscle weakness on the left (opposite side) unclear cause (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis bilateral (Musculoskeletal and connective tissue disorders) | 1 (1)
gonarthrosis left (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis on both sides of the lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis right (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis right , causes discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis right and left (Musculoskeletal and connective tissue disorders) | 1 (1)
Head pain due to back complaints (Musculoskeletal and connective tissue disorders) | 1 (1)
Heart failure DD: TAA (Cardiac disorders) | 1 (1)
Heart failure NYHA III (Cardiac disorders) | 1 (1)
Herniated Disc (Musculoskeletal and connective tissue disorders) | 1 (1)
herniated disc lumbar spine with stiffening (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes Zoster (previously known, now recurrence post-op) (Infections and infestations) | 1 (1)
Hip pain partly on right, partly on left, partly due to foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 10 (10)
Ignition of the other hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 2 (2)
Internal problems. Hips do not cause problems (General disorders) | 1 (1)
Jumping of the tractus ibiotibialis (coxa saltans) (Musculoskeletal and connective tissue disorders) | 1 (1)
Kidney insufficiency (Renal and urinary disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee pain left - no relationship to study device (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee problems (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee problems left side, age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee TEP left (Musculoskeletal and connective tissue disorders) | 1 (2)
Left hip (not study hip) pain, needs to be replaced (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip causes problems but no diagnosis available (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
left hip problems for 3 years (only medication) (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip TEP (non-study hip) still complaints, leg length difference due to TEP on the left (Musculoskeletal and connective tissue disorders) | 1 (1)
Limitation of walking distance (Musculoskeletal and connective tissue disorders) | 1 (1) — And only light physical activities due to hip TEP independent leg pain
Local swelling and redness with puncture without evidence of pathogens (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower leg wound after trauma (Skin and subcutaneous tissue disorders) | 1 (1)
Lumbar sciatica. Spinal canal sterosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spine complaints due to slight lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spine discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphedema bilateral varicosis (Cardiac disorders) | 1 (1)
Lymphoedema left leg 2017 (Cardiac disorders) | 1 (1)
Mild spinal stenosis of the lumbar spine- lumbar spine stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Mitral insufficiency (Cardiac disorders) | 2 (2)
Multiple herniated discs (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis ossificans (Musculoskeletal and connective tissue disorders) | 1 (1)
Nerve paralysis, siatic nerve lesion (Nervous system disorders) | 1 (1)
Nerve paralysis, weakness of the peroneus, already regressing at discharge (Nervous system disorders) | 1 (1)
Obstructive sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Occasional hip pain (study hip) (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis in large joints (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain both knees (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain from time to time in both knees (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in knee joint after knee TEP (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in the contralateral hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in the right groin (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain right knee, age-related not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Painkillers for back pain, spondylarthrosis herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Painkillers for pain in lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Feeling of uncertainty during walk (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle weakness in legs and joint pain in knees and ankle
Patient has back problems (Musculoskeletal and connective tissue disorders) | 1 (1)
Patient has had stomach problems (Gastrointestinal disorders) | 1 (1)
Patient slipped. 6 weeks groin pain right side, 03.08.2016-09.2016 (Musculoskeletal and connective tissue disorders) | 1 (1)
Patient was in general not very satisfied (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient often had the feeling that hip will "slip out".
pAVK right, reason for more pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Perioperative Anemia (Blood and lymphatic system disorders) | 10 (10)
Peripheral artery disease (Cardiac disorders) | 1 (1)
Phlebolymphedema (Cardiac disorders) | 1 (1)
Polyarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 3 (3)
Poor general condition, no relationship to study device (General disorders) | 1 (1)
Poor general condition. Patient with dementia. Polarstem in situ (Psychiatric disorders) | 1 (1)
Poor general health condition (General disorders) | 3 (4)
Poor general health condition, psychiatric disorders (Psychiatric disorders) | 1 (1)
Postoperative anemia (Blood and lymphatic system disorders) | 1 (1)
Pressure pain medial tibial head with knee prosthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Progressive complaints in various areas of Musculoskeletal & connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) — Degenerative cervical/lumbar spine syndrome, SI joint affection, gonarthrosis, impingment syndrome of the shoulders. No association with study procedure, Repeated analgesic therapy for
Pronounced coxarthrosis on the right (Musculoskeletal and connective tissue disorders) | 1 (1)
Prosthesis in situ. Patient reports minimal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pseudomembranous colitis (not related to study procedure) (Gastrointestinal disorders) | 1 (1)
Recurrent depressive disorder (Psychiatric disorders) | 1 (1)
Reflux (Gastrointestinal disorders) | 1 (1)
resection of a liver metastasis (Hepatobiliary disorders) | 1 (1)
Restless Leg Syndrom (Nervous system disorders) | 1 (1)
Right hip problems due to obesity and age-related. Not related to study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Right knee pain now and then (Musculoskeletal and connective tissue disorders) | 1 (1)
Right tronchanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rollator since 4 years due to MS (Nervous system disorders) | 1 (1)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p meniscuc lesion left 2017. No relation to study procedure (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p pericardial effusion (Cardiac disorders) | 1 (1)
s/p rotator cuff rupture left (Musculoskeletal and connective tissue disorders) | 1 (1)
s/p rotator cuff rupture right (Musculoskeletal and connective tissue disorders) | 1 (1)
Schmerzen in der Wirbelsaeule (Musculoskeletal and connective tissue disorders) | 1 (1)
Seroma drainage post-op (Musculoskeletal and connective tissue disorders) | 1 (1)
severe pain and swelling in right knee (Gonarthrosis) (Musculoskeletal and connective tissue disorders) | 1 (1)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1)
Since 4 months problems with spinal discs causing pain in non study hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Slight coxarthrosis on the left (non study hip) (Musculoskeletal and connective tissue disorders) | 1 (1)
Small intestine passage disorder (Gastrointestinal disorders) | 1 (1)
Spinal canal stenosis and thus back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal canal stenosis lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal canal stenosis of the cervical and lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylarthrosis lumbar spine (Musculoskeletal and connective tissue disorders) | 2 (2)
Spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiffening of contralateral hip joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Torn tendon on shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tricuspid insufficiency (Cardiac disorders) | 1 (1)
Tronchanteric bursitis (Musculoskeletal and connective tissue disorders) | 8 (8)
Upper abdominal complaints (Gastrointestinal disorders) | 1 (1)
Ureteritis (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Vitamin B12 deficiency (General disorders) | 1 (1)
Wobbly knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Wound dressing allergy (Immune system disorders) | 1 (1)
Z.n. Cerebral hemorrhage in 2008 with subsequent shunt implantation (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-11-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02648152/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02648152/SAP_001.pdf